CLINICAL TRIAL: NCT06412250
Title: A Prospective, Open-Label, Multi-Country, Multicentre, Observational PoSt Market SurvEillance of VIVO ISAR (Polymer-Free Sirolimus Eluting Coronary Stent System) In Real World Patients Undergoing PCI With Short Dual Antiplatelet Therapy
Brief Title: A Multicenter Observational Registry to Evaluate Safety and Performance of Vivo ISAR (SECURE Global Registry)
Status: Recruiting | Type: Observational
Sponsor: Translumina Therapeutics Pvt Ltd. (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: TL/SECURE/VIVO/2023-01
Record Dates: First submitted 2024-05-08; First posted 2024-05-14 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this post marketing observational registry is to evaluate clinical outcomes (safety and performance) in an all-comers population with coronary artery disease (CAD) treated with the Polymer Free Sirolimus Eluting Coronary Stent Vivo ISAR and planned for an abbreviated (≤ 3 months) dual antiplatelet therapy (DAPT) regimen.

DETAILED DESCRIPTION:
This study is a prospective, observational, multi-country, multi-Centre, single-arm registry designed to evaluate the clinical safety and performance of VIVO ISAR, Polymer Free Sirolimus Eluting Coronary Stent System. The study population is made up of subjects who have undergone PCI using VIVO ISAR and are receiving standard of care short DAPT treatment (≤ 3 months) . Subjects will be screened by site teams and offered the opportunity to participate in the registry after their procedure. Rationale for this study is to evaluate clinical outcomes and collect data of the Polymer Free Sirolimus Eluting Coronary Stent in real world CAD patients with follow-up at 1 month, 3 months and 12 months.

All medications and procedures to be used/ performed in this registry are commonly used/performed for clinical indications as part of standard of care and have well-defined safety profiles.

The study does not influence the choice of device utilized nor does it alter the routine standard of care. After a patient has been treated with the Vivo ISAR, informed consent will be requested and the eligible patient will be registered in the study.

Baseline data will be completed using medical notes. All recruited subjects will then be followed as per routine practice together with telephonic follow-up at 30 days, 3 months and 12 months from the baseline PCI procedure date.

The 30 day, 3 months and 12 month telephonic follow up will consist of a verbally report of the DAPT anticoagulation medications continued, about any lab assessments that might have happened, recording of any adverse events, and any interventional treatment that has occurred since previous contact.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent.
2. Treated only with the VIVO ISAR stent system.
3. ≥ 18 years old.
4. Male or non-pregnant female patient.
5. Intended for treatment with ≤ 3 months DAPT after PCI as per standard of care.

Exclusion Criteria:

1. Patients having any of the following conditions will not be considered (enrolled) for the study Concurrent participation in an interventional study.
2. Cardiogenic shock/hemodynamic instability around the time of the index procedure.
3. Concurrent medical condition with a life expectancy of less than 12 months.
4. Allergy or contraindication to antiplatelet therapy, cobalt chromium, sirolimus or any known hypersensitivity to the planned anti-platelet drugs.
5. History of cerebrovascular accident in the last 6 months.
6. Pregnant female.
7. PCI performed within the previous 3 months from the date of index procedure
8. Treated with another stent type during the index procedure in addition to the VIVO ISAR stent system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A real-world population undergoing percutaneous coronary intervention with VIVO-ISAR (Polymer Free Sirolimus Eluting Coronary Stent) and intended for treatment with ≤ 3 months of DAPT
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Ischemic endpoint | 12 months
  Cardiovascular death, myocardial infarction (not clearly attributable to a non-target vessel), definite or probable stent thrombosis or urgent target lesion revascularization (TLR).
Bleeding endpoint | 12 months
  bleeding defined as Bleeding Academic Research Consortium (BARC) class 3 or higher

SECONDARY OUTCOMES:
All-cause mortality | 12 months
  Mortality
Cardiovascular death | 12 months
  * Any death due to proximate cardiac cause (e.g., myocardial infarction, low-output failure, fatal arrhythmia).
  * Unwitnessed death and death of unknown cause.
  * All procedure-related deaths (including those related to concomitant treatment).
Myocardial infarction (MI) | 12 months
  Myocardial Infarction (including periprocedural myocardial infarction) as defined per the Fourth Universal Definition of Myocardial Infarction: "Detection of a rise and/or fall of cardiac troponin (cTn) with at least one value above the 99th percentile and with at least one of the following:
  1. Symptoms of acute myocardial ischemia;
  2. New ischemic electrocardiographic (ECG) changes;
  3. Development of pathological Q waves;
  4. Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality in a pattern consistent with an ischemic etiology;
  5. Identification of a coronary thrombus by angiography including intracoronary imaging or by autopsy."
Stroke | 12 months
  caused either by a clot obstructing the flow of blood to the brain (called an ischemic stroke) or by a blood vessel rupturing and preventing blood flow to the brain (called a hemorrhagic stroke)
Stent thrombosis (definite/probable) | 12 months
  Definite Stent Thrombosis:
  Angiographic confirmation of stent thrombosis:
  * The presence of a thrombus that originates in the stent or in the segment 5 mm proximal or distal to the stent and presence of at least one of the following criteria within a 48-hour time window:
  * Acute onset of ischemic symptoms at rest
  * New ischemic ECG changes that suggest acute ischemia
  * Typical rise and fall in cardiac biomarkers
    b) Probable Stent Thrombosis Clinical definition of probable stent thrombosis is considered to have occurred after intracoronary stenting in the following cases:
  * Any unexplained death within the first 30 days.
  * Irrespective of the time after the index procedure, any MI that is related to documented ischemia in the territory of the implanted stent without angiographic confirmation of stent thrombosis and in the absence of any other obvious cause.
Target Lesion Revascularisation (TLR) - Ischemia driven (ID) | 12 months
  A TLR is considered ischemia-driven if angiography at follow-up shows a percent diameter stenosis ≥50% and if one of the following occurs:
  * Positive history of recurrent angina pectoris, presumably related to the target vessel.
  * Objective signs of ischemia at rest (ECG changes) or during exercise test (or equivalent), presumably related to the target vessel.
  * Abnormal results of any invasive functional diagnostic test (e.g., Doppler flow velocity reserve, fractional flow reserve).
  * A target lesion revascularisation (TLR) or target vessel revascularisation (TVR) with a diameter stenosis ≥70% even in the absence of the above-mentioned ischemic signs or symptoms TLR events which do not meet the criteria for ID-TLR are considered non-ID TLR events
Urgent TLR | 12 months
  Acute condition post index procedure where urgent revascularization of the target lesion is necessary
Target vessel revascularisation (TVR) | 12 months
  repeat percutaneous intervention or surgical bypass of any segment of a target vessel.
BARC class 2 bleeding | 12 months
  any overt, actionable sign of hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Prof Adnan Kastrati, Study Chair — German Heart Centre Munich, Germany; Prof Azfar Zaman, Principal Investigator — Freeman Hospital, Newcastle, UK
Locations (31):
- India (16):
  - Zydus Hospitals, Ahmedabad
  - Fortis Hospital, Bangalore
  - Adesh Hospital, Bathinda
  - PGIMER, Chandigarh
  - National Heart Institute, Delhi
  - Fortis Escorts Heart Institute & Research Centre, Delhi
  - Medanta-The Medicity, Gurugram
  - Yashoda Hospitals, Hyderabad
  - Shalby Hospital, Jabalpur
  - Fortis Hospital, Kalyān
  - L.P.S Institute of Cardiology, Kanpur
  - Fortis Hospital, Kolkata
  - Dr. Ram Manohar Lohia Hospital (RML), Lucknow
  - Seva Sadan Hospital, Miraj
  - Fortis, Mohali
  - Yashodha Hospital, Somājigūda
- Italy (7):
  - ASREM - Regional Hospitals, Campobasso
  - Montevergine, Mercogliano AV
  - Clinica Mediterranea, Napoli
  - University of Padua, Padova, Padua
  - Clinica Pierangeli, Pescara
  - Santo Spirito Hospital, Pescara
  - Tor Vergata University, Roma
- Netherlands (3):
  - Amsterdam UMC (University Medical Centers), Amsterdam
  - Tergooi MC, Hilversum
  - Viecuri MC, Venlo
- United Kingdom (5):
  - Bedford Hospital, Bedford
  - Freeman Hospital, Newcastle
  - Derriford Hospitalm Plymouth NHS Trust, Plymouth
  - Salisbury NHS Foundation Trust, Salisbury
  - Wrightington, Wigan and Leigh Teaching Hospitals NHS Foundation Trust, Wigan

IPD SHARING:
Plan to Share IPD: No